CLINICAL TRIAL: NCT01252277
Title: Modulation of Breast Cancer Risk Biomarkers in Premenopausal Women by High Dose Omega-3 Fatty Acids
Brief Title: Breast Cancer Risk Biomarkers in Premenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Carol Fabian, MD (Other)
Responsible Party: Sponsor-Investigator, Carol Fabian, MD, Professor, Director Breast Cancer Prevention Unit, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 12349
Record Dates: First submitted 2010-11-23; First posted 2010-12-02 (Estimated); Results first posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lovaza™ (Experimental): Lovaza™ (two 1 gram capsules twice daily) for six months
  Interventions: Drug: Lovaza™

INTERVENTIONS:
Drug: Lovaza™ — 4 capsules daily for 6 months
  Other Names: esters of EPA and DHA

SUMMARY:
This study is designed to gather information on how the prescription drug Lovaza™ which contains omega-3 fatty acids, affects blood and tissue risk biomarkers for breast cancer. This drug is currently approved by the FDA for reducing blood levels of triglycerides.

DETAILED DESCRIPTION:
The central hypothesis is that 6 months of administration of high dose omega-3 fatty acid esters [eicosapentaenoic acid (EPA) 1860 mg, and docosahexaenoic acid (DHA) 1500 mg] daily in the form of a standard prescription strength dose of Lovaza™ (two 1 gram capsules twice daily) will have a favorable side effect profile and potential efficacy as demonstrated by favorable modulation of one or more blood and breast tissue risk biomarkers for breast cancer in premenopausal women.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be premenopausal and between the ages of 25 and 54 and must have had a menstrual period within the past 12 months. Women who are not menstruating regularly due to use of certain types of contraceptives may be entered with restrictions. Their estrogen progesterone, and follicle stimulating hormone (FSH) levels must be documented at baseline random periareolar fine needle aspiration (RPFNA) and their off study RPFNA must take place at a similar portion of their cycle (high or low progesterone levels). In order to do this a serum progesterone will have to be obtained ~ 4 weeks before planned RPFNA and again 2 weeks later such that the RPFNA can be performed in the same phase of the "cycle" as baseline.
* Subjects must be at increased risk for breast cancer on the basis of at least one of the following criteria:
* A five-year Gail risk of ≥ 1.67% or three times the average risk for a woman of the same age using either the Surveillance Epidemiology and End Results (SEER, http://seer.cancer.gov) database or the NCI Breast Cancer Risk Assessment Tool (www.cancer.gov/bcrisktool)., or 10 yr Tyrer-Cuzick risk twice that of the population risk as listed in model, or RPFNA atypia
* BMI <40 Kg/m3
* A first degree relative with breast cancer under the age of 60 or multiple second degree relatives with breast cancer.
* Multiple prior biopsies or at least one prior biopsy exhibiting atypical hyperplasia (AH), lobular carcinoma in situ (LCIS), ductal carcinoma in situ (DCIS).
* RPFNA evidence of hyperplasia with atypia within the last three years;
* Chest or neck radiation before age 30;
* Mammographic breast density by visual estimate equals or exceeds 50%.
* Subjects must be willing to continue the same hormonal milieu present at baseline throughout trial. If not using an oral, vaginal, or topical contraceptive, must be willing to actively use barrier methods of contraception to prevent pregnancy.
* Six months or more must have elapsed from completion of a prevention intervention trial (with exception of a weight reduction trial), ingestion of a selective estrogen receptor modulator (SERM) or aromatase inhibitor (AI) prior to baseline biomarker assessment.
* Subjects must be willing to undergo measurement of height, weight, and BMI and undergo body composite analysis (DEXA) at initiation and conclusion of intervention.
* Subjects with a history of AH, LCIS, or ER-positive DCIS by diagnostic biopsy, must have been counseled about appropriate standard prevention therapies such as tamoxifen and are either not eligible or are not interested in standard prevention therapies. Women with DCIS must have had appropriate local therapy (lumpectomy plus radiation or mastectomy). If subject has had a DCIS, at least two months must have elapsed from surgery and/or radiation therapy to the involved breast. Only the contralateral (uninvolved breast) will be studied by RPFNA. The subject may not have had any radiation therapy to the contralateral breast to be studied
* Subjects > 40 must have had a screening mammogram within 6 months of entering the interventional portion of the study and read as not suspicious for breast cancer or if suspicious must have completed all suggested tests including biopsy and found to have no evidence of cancer. Subjects of sufficient age and/or risk for a baseline mammogram must be willing to have an off-study mammogram performed 6 months after study entry.
* Subjects must have had an RPFNA of the breast within six months prior to entering the intervention portion of the study and be willing to have another RPFNA at ~6.5 months after starting Lovaza™.
* Tissue Eligibility: Subjects must have cytomorphologic evidence of hyperplasia with atypia or borderline atypia (Masood score 14 or higher). There must be ≥500 epithelial cells on the slide for cytomorphology and evidence of proliferation by Ki-67 staining. There must be sufficient reserved methanol- formalin-fixed material for real time quantitative polymerase chain reaction (RT-qPCR). Frozen tissue must also have been obtained for fatty acid analysis, reverse phase proteomics, adipokines and cytokines, and RT-qPCR.
* Subjects must be willing to undergo phlebotomy at baseline, and 6 months and 6.5 months approximately 3 tablespoons of blood will be obtained at baseline, and 6 months and 6.5 months or 6 tablespoons if the subject decides to participate in the optional monocyte cytokine release assay .
* Subjects must produce a spot urine sample at baseline, 6 months and at study conclusion. Baseline urine sample will in part be used to document that subject is not pregnant.
* Subjects must be willing to complete questionnaires regarding diet and supplement use, quality of life, relevant family history, personal health and reproductive history and medications at initiation and conclusion of the intervention.
* Subjects must be willing to sign an informed consent for the entire study and separate consent for repeat RPFNA

Exclusion Criteria

* Women that have had a metastatic malignancy of any kind.
* Women that have had prior invasive breast cancer, diagnosed or treated within the past five years.
* Women who are currently taking anticoagulants.
* Women who have breast implants.
* Women who have undergone change in their hormonal milieu in the past 6 months this includes pregnancy, lactation, or stopping or starting hormonal contraceptives..
* Women who have taken omega 3 fatty acid supplements within 3 weeks prior to their baseline RPFNA.
* Women who regularly take NSAIDS (>7 tablets weekly).

Inclusion of Women and Minorities

-This study utilizes women at increased risk for breast cancer. Subjects recruited from an established cohort of women followed in the Breast Cancer Prevention Center. From previous trials we can expect 6% minority accrual which is similar to our hospital demographics. Males are not included due to the low absolute risk of breast cancer, and the difficulty of performing RPFNA on the male breast.

Ages: 25 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2010-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women at high risk for development of breast cancer, seen in the Breast Cancer Prevention Center at the University of Kansas Medical Center.
  Recruitment December 2010 to August 2012
Groups:
- Lovaza™: Lovaza™: 4 capsules (total of 1860 mg EPA + 1500 mg DHA) daily for 6 months
Period: Overall Study
Arm/Group | Lovaza™
Started | 36
Completed | 34
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lovaza™
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.9 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
Gail 5-year Projected Probability of developing breast cancer [Mean (Standard Deviation); unit: Projected Probability, percent] | 2.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects That Complete an Intervention of Lovaza™ 4 Grams Per Day
Description: The proportion of subjects that complete an intervention of Lovaza™ 4 grams per day (~ 1800 mg EPA and 1500 mg DHA) administered for 6 months to premenopausal women under age 55.
Time Frame: 6 month visit
Measure: Number; unit: proportion of enrolled participants
Arm/Group | Lovaza™
Number analyzed (Participants) | 36
proportion of enrolled participants | 0.94

2. Secondary Outcome: Modulation of the Risk Biomarker Masood Score
Description: Change in the semiquantitative cytology index score (Masood score) from baseline to end of study. Masood Score range 6 - 24; increasing values denote increasing cytologic abnormality. Thus, negative values for change reflect an improvement, i.e., less cytologic abnormality after intervention.
Time Frame: 6 month value compared to baseline value
Measure: Median (Inter-Quartile Range); unit: change in units on a scale
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
change in units on a scale | -1 [-3 to 0]
Statistical Analysis 1: Comparison: Lovaza™; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance, p<0.05

3. Secondary Outcome: Modulation of Ki-67 Expression
Description: Change (baseline to end of study) in percent of benign breast epithelial cells exhibiting immunostaining for Ki-67
Time Frame: 6 month value compared to baseline value
Measure: Median (Inter-Quartile Range); unit: Change in percent Ki-67 expression
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
Change in percent Ki-67 expression | -1.45 [-2.55 to 0]
Statistical Analysis 1: Comparison: Lovaza™; Test type: Superiority or Other; p = 0.021, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons

4. Secondary Outcome: Change in (DHA+EPA):AA Ratio for Phospholipids in Plasma.
Description: Change (from baseline to end of study) for the ratio derived from levels of DHA, EPA, and Arachadonic Acid (AA); measured as percent of total fatty acid content in the phospholipid compartment of plasma.
Time Frame: baseline to end of intervention (~6 months)
Population: Subjects completing intervention
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
ratio | 0.61 [0.34 to 0.81]
Statistical Analysis 1: Comparison: Lovaza™; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance p<0.05

5. Secondary Outcome: Change in Quality of Life.
Description: Change in score on Breast Cancer Prevention Trial (BCPT) Symptom Checklist. 43 symptoms, each scored as 0 to 4, are summed to provide a global score (range 0 to 172). Increasing score represents increasing problems with side effects. For change in score over period of intervention, a negative score indicates an improvement in quality of life while a positive score indicates increasing interference with daily activities due to worsening symptoms. Theoretically, the range of change could be -172 to +172.
Time Frame: duration of intervention, baseline to ~ 6 months
Population: Subjects completing intervention
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Lovaza™
Number analyzed (Participants) | 34
units on a scale | 1.0 [-2.25 to 3.0]
Statistical Analysis 1: Comparison: Lovaza™; Test type: Superiority or Other; p = 0.48, Wilcoxon (Mann-Whitney) — No adjustment for multiple comparisons. A priori threshold for statistical significance, p<0.05

ADVERSE EVENTS:
Time Frame: duration of intervention, planned at 6 months
Arm/Group | Lovaza™
Serious Adverse Events (participants affected / at risk) | 0/36
Other Adverse Events (participants affected / at risk) | 25/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lovaza™ (N=36)
Headaches (Nervous system disorders) | 13 (13)
increased bilirubin (Metabolism and nutrition disorders) | 2 (2)
Hot flashes (Endocrine disorders) | 2 (2)
breast tenderness or sensitivity (Reproductive system and breast disorders) | 3 (3)
joint pains (Musculoskeletal and connective tissue disorders) | 3 (3)
early awakening (Nervous system disorders) | 2 (2)
short temper (Psychiatric disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes